CLINICAL TRIAL: NCT00059462
Title: Phase I/II Randomized, Double Blind, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Subcutaneous Bay 50-4798 Administration in Patients With HIV Infection on Highly Active Antiretroviral Therapy (HAART) Compared to Patients on HAART Alone.
Brief Title: Safety and Efficacy of BAY 50-4798 in Patients With HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10630; NCT00048191 (obsolete NCT alias)
Record Dates: First submitted 2003-04-25; First posted 2003-06-02 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infections
Keywords: Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Interleukin-2 SA
- Arm 2 (Active Comparator)
  Interventions: Drug: HAART

INTERVENTIONS:
Drug: Interleukin-2 SA — HAART and Bay 50-4798
  Arms: Arm 1
Drug: HAART — HAART alone
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the safety of the experimental drug Bay 50-4798 in HIV positive patients receiving HAART and to test the drug's effect on the CD4+ T-cell count.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection (positive enzyme linked immuno assay (EIA) confirmed by Western Blot).
* Age greater than or equal to 18 years.
* Plasma HIV viral load less than 10,000 copies/ml (by bDNA assay or less than 14,000 copies/ml by RT-PCR) on at least 2 occasions within 8 weeks prior to study entry with no more than a 0.5 log increase between the most recent and the earlier viral load measurements.
* CD4 + T-cell count greater than or equal to 200/mm(3) on at least 2 occasions within 8 weeks of study entry.
* On a stable HAART regimen for greater than or equal to 8 weeks.
* Karnofsky Score greater than or equal to 80.
* Written informed consent. Exclusion Criteria:
* Prior treatment with IL-2 or an IL-2 analogue.
* Pregnancy or breastfeeding. - Use of any known immunomodulators, cytokines, growth factors or systemic corticosteroids (e.g. prednisone greater than or equal to 15 mg/day or equivalent) within 4 weeks prior to study enrollment.
* History of an AIDS defining illness by the Centers for Disease Control (CDC) definition within 8 weeks prior to study entry.
* Acute bacterial or viral infection within 4 weeks prior to enrollment.
* Received an immunization within 4 weeks prior to enrollment.
* History of autoimmune disease including psoriasis, inflammatory bowel disease.
* Medical history of transplantation (solid organ or bone marrow).
* Received an investigational drug in the past 30 days other than Food and Drug Administration (FDA) sanctioned treatment IND antiretroviral agents.
* Renal insufficiency with a serum creatinine level greater than 1.5 times the upper limit of normal.
* Bone marrow suppression as defined by one or more of the following: granulocyte count less than 1,000 cells/ÂµL; hemoglobin less than 9.0g (females) or less than 9.5g (males); or platelet count less than 75,000 cells/ÂµL.
* Evidence of hepatic disease indicated by one or more of the following: SGOT (AST) and/or SGPT (ALT) greater than 5 times the upper limit of normal. Bilirubin greater than 2 times the upper limit of normal (except for patients with known Gilbert's syndrome or those receiving indinavir who may be enrolled if the serum bilirubin is less than or equal to 5 times the upper limit of normal).
* Active cardiac disease (coronary artery disease, congestive heart failure or cardiomyopathy) requiring treatment with any of the following medications: antiarrhythmic agents including digitalis, anti-anginal drugs including topical or systemic nitrates, calcium channel blockers, and beta blockers, and afterload reducers including ACE inhibitors. Patients requiring any of these medications solely for the treatment of hypertension remain eligible for the study.
* Presence of significant cardiac insufficiency (greater than or equal to New York Heart Association Grade 2).
* Diagnosis of an active malignancy requiring treatment with systemic cytotoxic chemotherapy.
* Active alcohol or substance abuse which, in the opinion of the investigator, will seriously compromise the subject's ability to adhere with the demands of the study.
* Any central nervous system (CNS) disease that requires active treatment with anticonvulsants.
* Use of an antimetabolite such as hydroxyurea within 4 weeks prior to study entry.
* Known co-infection with Hepatitis B or C virus unless serum transaminases are less than or equal to 2 times the upper limit of normal on at least two occasions within 8 weeks prior to study entry.
* Known CD4 Nadir less than 50 cells/mm(3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- United States (8):
  - Birmingham, Alabama
  - Davis, California
  - Los Angeles, California
  - Palo Alto, California
  - San Francisco, California
  - Chicago, Illinois
  - Bethesda, Maryland
  - Cleveland, Ohio
- Créteil, France
- London, Greater London, United Kingdom